CLINICAL TRIAL: NCT06976619
Title: The Effect of Glycemic Control and of GLP-1 Receptor Agonism on Islet GLP-1 in People
Brief Title: The Effect of Glycemic Control and of GLP-1 Receptor Agonism on Islet GLP-1 in People With Type 1 and Type 2 Diabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 24-007682
Record Dates: First submitted 2025-05-05; First posted 2025-05-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Islet Function; Glucose Toxicity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant
Masking Description: Intervention will be assigned in single-blind fashion (Placebo pens for liraglutide are unavailable). A placebo syringe created by Research Pharmacy in addition to 'masked' liraglutide pens will be used over 4-weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Type 1 diabetes - Placebo arm (Placebo Comparator): Subjects will receive syringes loaded with saline to self-administer daily during the intervention phase
  Interventions: Other: Saline Injections
- Type 1 diabetes - Liraglutide arm (Active Comparator): Subjects will receive 0.6mg Liraglutide syringes to self-administer daily during the intervention phase
  Interventions: Drug: Liraglutide Pen Injector
- Type 2 diabetes - Placebo arm (Placebo Comparator): Subjects will receive syringes loaded with saline to self-administer daily during the intervention phase
  Interventions: Other: Saline Injections
- Type 2 diabetes - Liraglutide arm (Active Comparator): Subjects will receive 0.6mg Liraglutide syringes to self-administer daily during the intervention phase
  Interventions: Drug: Liraglutide Pen Injector

INTERVENTIONS:
Drug: Liraglutide Pen Injector — Liraglutide 0.6mg
  Other Names: Liraglutide
  Arms: Type 1 diabetes - Liraglutide arm; Type 2 diabetes - Liraglutide arm
Other: Saline Injections — Saline in syringes to serve as placebo for single blind study
  Other Names: Placebo
  Arms: Type 1 diabetes - Placebo arm; Type 2 diabetes - Placebo arm

SUMMARY:
The investigators recently demonstrated that blockade of Glucagon-Like Peptide-1's (GLP-1) receptor (GLP1R) results in changes in islet function without changes in circulating GLP-1. These effects are more pronounced in people with early type 2 diabetes (T2DM) in keeping with increased expression of PC-1/3 and GLP-1 that is observed in diabetic islets. However, its regulation is at present unknown. There is evidence that α-cell proglucagon processing is subject to paracrine regulation by the β-cell3. It is unclear if the effects of GLP1R agonism on islet GLP-1 differ in Type 1 diabetes (T1DM) compared to T2DM. This experiment will examine the effect of glycemic control ± a GLP1R agonist on islet GLP-1 in people with (T2DM) and without (T1DM) β-cells.

DETAILED DESCRIPTION:
The investigators recently demonstrated that blockade of Glucagon-Like Peptide-1's (GLP-1) receptor (GLP1R) results in changes in islet function without changes in circulating GLP-1. This supports other evidence (rodents and humans) that through the (inducible) expression of a prohormone convertase (PC-1/3), the α-cell can process proglucagon to intact GLP-15,6. 'Islet' or 'pancreatic' GLP-1 acts in a paracrine fashion to regulate insulin (basal and 1st phase) and glucagon secretion. These effects are more pronounced in people with early type 2 diabetes (T2DM) in keeping with increased expression of PC-1/3 and GLP-1 that is observed in diabetic islets.

There is evidence that α-cell proglucagon processing is subject to paracrine regulation by the β-cell. β-cell secretion of the signaling peptide 14-3-3-Zeta is decreased by GLP1R agonism (Fig.1), stimulating α-cell production of GLP-1. This is a testable hypothesis in humans; people with type 1 diabetes (T1DM) have dysregulated glucagon secretion and evidence of islet GLP-1. It is unclear if the effects of GLP1R agonism on islet GLP-1 differ compared to T2DM. This experiment will examine the effect of glycemic control ± a GLP1R agonist on islet GLP-1 in people with (T2DM) and without (T1DM) β-cells.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes treated with insulin

Exclusion Criteria:

1. Age < 25 or > 70 years.
2. HbA1c > 10.0%
3. For female subjects: positive pregnancy test at the time of enrollment or study
4. History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
5. Prior use of GLP-1 receptor agonists in the previous year.
6. Active systemic illness or malignancy.
7. Symptomatic macrovascular or microvascular disease.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of exendin 9-39 on fasting glucagon secretion rate before and after liraglutide treatment | The change in fasting glucagon secretion rate (saline vs. exendin 9-39) in the baseline study will be compared with the change in fasting glucagon secretion rate (saline vs. exendin 9-39) after 30 days of treatment with liraglutide (post-liraglutide)
  Glucagon secretion rate will be estimated by deconvolution from glucagon concentrations during fasting (-30 to 0 min) of each study day.
Effect of exendin 9-39 on glucagon secretion rate during hyperglycemia before and after liraglutide | The change in glucagon secretion rate during hyperglycemia (saline vs. exendin 9-39) in the baseline study will be compared with the change (saline vs. exendin 9-39) after 30 days of treatment with liraglutide (post-liraglutide)
  Glucagon secretion rate will be estimated by deconvolution from glucagon concentrations during hyperglycemia (150 to 180 min) of each study day.

SECONDARY OUTCOMES:
Effect of exendin 9-39 on fasting glucagon secretion rate in people with type 1 diabetes vs type 2 diabetes | The change in fasting glucagon secretion (saline vs. exendin 9-39) in the baseline studies will be compared in people with type 1 diabetes vs type 2 diabetes
  Glucagon secretion rate will be estimated by deconvolution from glucagon concentrations during fasting (-30 to 0 minutes) during the baseline studies
Effect of exendin 9-39 on glucagon secretion rate during hyperglycemia in people with type 1 diabetes vs type 2 diabetes | The change in glucagon secretion during hyperglycemia (saline vs. exendin 9-39) in the baseline studies will be compared in people with type 1 diabetes vs type 2 diabetes
  Glucagon secretion rate will be estimated by deconvolution from glucagon concentrations during hyperglycemia (150 to 180 minutes) during the baseline studies

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No